CLINICAL TRIAL: NCT06220071
Title: Retrospective Multicentric European Study In Patients With Vertebral Metastases (Train-Metastra)
Brief Title: Multicentric European Study In Patients With Vertebral Metastases
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: Train-METASTRA
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Spinal Metastases
Keywords: risk of fracture; spinal instability; decision support system; artificial intelligence-based models; mechanistic personalised model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vertebral metastases: Patients affected by spinal metastases that are not surgically treated
  Interventions: Other: Case series review of clinical and radiographic data

INTERVENTIONS:
Other: Case series review of clinical and radiographic data — Extraction of clinical and radiographic data related to patients' history from medical records

SUMMARY:
Train-METASTRA is a retrospective study that will be performed in order to collect a large and harmonised amount of clinical and imaging data concerning vertebral metastases, focusing in particular on the risk of fractures. This type of dataset will be created from the medical records of 2000 patients admitted in the last ten years in the four European clinical centers participating in METASTRA project: "COMPUTER-AIDED EFFECTIVE FRACTURE RISK STRATIFICATION OF PATIENTS WITH VERTEBRAL METASTASES FOR PERSONALISED TREATMENT THROUGH ROBUST COMPUTATIONAL MODELS VALIDATED IN CLINICAL SETTINGS", funded by the European Union under the call "HORIZON-HLTH-2022-TOOL-12-two-stage/Computational models for new patient stratification strategies". The project is coordinated by the University of Bologna (UNIBO) (PI prof. Luca Cristofolini) and involves 15 European partners, including Sarl Voisin Consulting Life Sciences VCLS, University of Szeged (Hungary), University of Sheffield (UK) and FrontEndART (Hungary).

This type of dataset is not currently available in the literature and it will be pivotal to the development of the METASTRA computational models for the stratification of the risk of fracture of patients affected by spinal metastases.

ELIGIBILITY:
Inclusion Criteria:

* Alive or dead
* Age 18 -99 years old
* Both male and female
* Diagnosis of cancer metastases at the spine
* Any SINS score
* Admitted for hospitalisation or outpatient visit from Jan 2012 to Dec 2022 N ≥ 1 non-stabilised metastatic vertebra
* Presence of baseline CT scan, and/or MRI and x-rays, showing the presence of metastatic lesions that are not surgically treated
* At least one follow-up visit at ≥ 3 months after the first evaluation or treatment

Exclusion Criteria:

* Minor patients
* Patients with diagnosis of primary spine tumour, degenerative spinal diseases, deformity or trauma
* Patients without non-stabilised vertebral metastases
* Patients without baseline CT scan or MRI
* Patients without follow up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The expected study population is a cohort of patients affected by spinal metastases admitted in the last ten years (from 2012 to 2022) in the four clinical centers involved in the study. This cohort of patients is characterised by the presence of one or more vertebral metastatic lesions that are not surgically treated.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
risk factors for vertebral fracture | at the baseline
  The primary objective of the study is to identify the main relevant characteristics to be used for stratifying the patients with vertebral metastases based on their risk of fracture.
risk factors for vertebral fracture | through study completion, an average of 1 year
  The primary objective of the study is to identify the main relevant demographic, clinical and radiographic characteristics to be used for stratifying the patients with vertebral metastases based on their risk of fracture.

SECONDARY OUTCOMES:
Critical metastases | after 1 year
  To classify critical metastases
AI-based models | after 1 year
  To train the data-driven computational models (METASTRA-AI) developed within the project
Physiology-based biomechanical models | after 1 year
  To inform the physiology-based biomechanical models (METASTRA-VPH) developed within the project

CONTACTS AND LOCATIONS:
Locations (3):
- Charite - Universitaetsmedizin Berlin, Berlin, Germany
- Budai Egeszsegkozpont Zrt, Budapest, Hungary
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes